CLINICAL TRIAL: NCT04673955
Title: Encorafenib and Cetuximab in Patients With Metastatic, BRAFV600E-mutated, Colorectal Carcinoma: a Multi-centric, Multi-national, Prospective, Longitudinal, Non-interventional Study in Germany, Austria and Switzerland
Brief Title: BRAF Inhibitor Encorafenib And Cetuximab Real Life Investigation of Next Generation CRC Treatment
Acronym: BERING-CRC
Status: Recruiting | Type: Observational
Sponsor: Pierre Fabre Pharma GmbH (Industry)
Collaborators: iOMEDICO AG (Industry); Pierre Fabre Pharma AG (Industry); Pierre Fabre Pharma Austria (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIS-PFO-2020-3101
Record Dates: First submitted 2020-10-08; First posted 2020-12-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Colorectal Carcinoma
Keywords: BRAFV600E mutation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Encorafenib — Observation of real-life treatment with encorafenib and cetuximab
  Other Names: Braftovi
Drug: Cetuximab — Observation of real-life treatment with encorafenib and cetuximab
  Other Names: Erbitux

SUMMARY:
The presence of a BRAFV600E mutation is a marker of poor prognosis in patients with mCRC and associated with a median overall survival (mOS) of approximately 12 to 14 months compared to 20 to 25 months for patients with BRAF wild-type tumours. After 1st line therapy, treatment outcomes with standard therapy are poor in patients with BRAF-mutated mCRC, with response rates (ORR) of ≤ 11%, a median progression-free survival (mPFS) between 1.8 and 2.8 months, and a mOS between 4.1 and 6.2 months. Failure to achieve adequate survival outcomes with standard treatment regimens in patients with BRAF-mutated mCRC has encouraged efforts to combine multiple targeted therapies: With 665 randomized patients, the BEACON CRC trial represents the largest trial and is currently the only phase III study in patients with BRAFV600E-mutant mCRC.

BERING CRC - designed as a prospective (allowing initial retrospective documentation), longitudinal, non-interventional study - will investigate the real-world effectiveness, quality of life, safety and tolerability of encorafenib and cetuximab in BRAFV600E-mutant mCRC patients, who have received prior systemic therapy. Data from this study will contribute to a deeper understanding and characterization to the everyday use of encorafenib and cetuximab in a broader patient population in the German, Austrian, and Swiss routine setting.

DETAILED DESCRIPTION:
The presence of a BRAFV600E mutation is a marker of poor prognosis in patients with mCRC and associated with a median overall survival (mOS) of approximately 12 to 14 months compared to 20 to 25 months for pa-tients with BRAF wild-type tumors. After 1st line therapy, treatment out-comes with standard therapy are poor in patients with BRAF-mutated mCRC, with response rates (ORR) of ≤ 11%, a median progression-free survival (mPFS) between 1.8 and 2.8 months, and a mOS between 4.1 and 6.2 months.

Failure to achieve adequate survival outcomes with standard treatment regimens in patients with BRAF-mutated mCRC has encouraged efforts to combine multiple targeted therapies: With 665 randomized patients, the BEACON CRC trial represents the largest trial and is currently the only phase III study in patients with BRAFV600E-mutant mCRC. After a safety lead in for dose confirmation of the triplet regimen, the phase III part was per-formed with a total of 665 patients, randomized 1:1:1 to either receive encorafenib plus binimetinib and cetuximab (triplet) or encorafenib plus cetuximab (doublet) or FOLFIRI / IRI plus cetuximab (control).

The BEACON CRC study met its primary endpoints Overall Response Rate (ORR) and Overall Survival (OS) comparing Encorafenib + Binimetinib + Cetuximab vs. Chemotherapy + Cetuximab (ORR: 26 vs. 2%, p<0.001; OS: median 9.0 vs. 5.4 months, HR 0.52, p<0.001). The BEACON CRC study was alpha-controlled also for the secondary endpoint comparing Encorafenib + Cetuximab vs. Chemotherapy + Cetuximab in terms of ORR and OS and showed a statistically significant advantage (ORR: 20 vs. 2%, p<0.001; OS: median 8.4 vs. 5.4 months, HR 0.60, p<0.001). In terms of safety, the overall frequency of adverse events grade 3/4 was 58% (En-corafenib + Binimetinib + Cetuximab) vs. 50% (Encorafenib + Cetuximab) vs. 61% (Chemotherapy + Cetuximab). Analysis of Quality of Life data resulted in a longer maintenance of Quality of Life in the Encorafenib + Binimetinib + Cetuximab arm and the Encorafenib + Cetuximab arm com-pared to Chemotherapy + Cetuximab. Between Encorafenib + Binimetinib + Cetuximab and Encorafenib + Cetuximab, no relevant differences were reported. With a longer Follow-Up (12.8 months) the updated OS data showed a median OS of 9.3 months in both the Encorafenib + Binimetinib + Cetuximab arm and the Encorafenib + Cetuximab arm compared to 5.9 months in the control arm. Updated ORR rates were 27% in the triplet arm (p<0.0001 vs. control), 20% in the doublet arm (p<0.0001 vs. control) and 2% in the control arm. The safety and tolerability were adequate, manage-able and consistent with the known profiles of BRAF-, MEK-, and EGFR-inhibitors. Regarding the triplet combination, the most common adverse events of any grade were diarrhea (triplet: 62%; control: 48%), dermatitis acneiform (triplet: 49%; control: 39%), nausea (triplet: 45%; control: 41%), and vomiting (triplet: 38%; control: 29%). Regarding the doublet combina-tion, the most common adverse events of any grade were nausea (34%), diarrhea (33%), fatigue (doublet 30%; triplet 33%; control 27%) and derma-titis acneiform (29%).

The most common updated grade ≥3 adverse events regarding the triplet combination were diarrhea (triplet: 11%; control: 10%), abdominal pain (triplet: 6%; control: 5%), nausea (triplet: 5%; control: 2%,vomiting (triplet: 5%; control: 3%) and intestinal obstruction (triplet 5%; control 3%). With the doublet regimen, the most common updated grade ≥3 adverse events were intestinal obstruction (doublet 5%), asthenia (doublet 4%; triplet 4%; control 5%), fatigue (doublet 4%; triplet 2%; control 5%), diarrhea (3%) and abdominal pain (3%).

Based on these data, it is expected that the European Medicines Agency (EMA) will approve encorafenib plus cetuximab for the treatment of adult patients with metastatic BRAFV600E-mutant CRC, who have received prior systemic therapy.

Data from pivotal clinical trials are usually based on a selected patient population in order to provide standardized results in the given indication. However, after marketing authorization usage in a broader patient popula-tion is to be expected. Therefore, BERINGCRC - designed as a prospective (allowing initial retrospective documentation), longitudinal, non-interventional study - will investigate the real-world effectiveness, quality of life, safety and tolerability of encorafenib and cetuximab in BRAFV600E-mutant mCRC patients, who have received prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient with regard to the pseudonymized documentation of his/her data in the frame of this non-interventional study
* Legally capable patient ≥ 18 years of age (no upper limit)
* Metastatic colorectal carcinoma with BRAFV600E-mutation, pretreated with systemic therapy
* Decision was taken to treat the patient with the doublet therapy (encorafenib and cetuximab) in accordance with the current SmPC and by prescription; this decision was taken prior to and independent from the inclusion into the study;
* Treatment with the doublet therapy (encorafenib plus cetuximab) has been started ≤ 3 months prior to providing written informed consent for this study or is planned to be started in the near future.

Exclusion Criteria:

* More than 2 prior systemic regimens in the metastatic setting (adjuvant systemic therapy with relapse ≤ 6 months will be counted as metastatic treatment line; maintenance treatment will not be counted as separate metastatic treatment line)
* Prior treatment with any RAF-inhibitor or MEK-inhibitor.
* Presence of any contraindication with regard to the doublet therapy (encorafenib plus cetuximab) as specified in the corresponding SmPCs
* Current or upcoming participation in an interventional clinical trial
* Current or upcoming systemic treatment of any other tumor than metastatic colorectal carcinoma
* Prisoners or persons who are compulsorily detained (involuntarily incarcerated).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic, BRAFV600E-mutant, colorectal carcinoma, who have received prior systemic therapy, with the decision to receive the doublet therapy encorafenib plus cetuximab according to the current SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | At 12 months after start of treatment
  Overall Survival rate

SECONDARY OUTCOMES:
Patient and disease profiles at start of treatment with encorafenib plus cetuximab | Baseline
  Demographic and disease chracteristics
BRAF-mutation assessment | Baseline
  Date and type of BRAFV600E testing
Type and sequence of treatments before and after encorafenib plus cetuximab | Through study completion, an average of 17 months
  Treatment sequence prior to and after encorafenib plus cetuximab
Characteristics of treatment with encorafenib plus cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Evaluation of reason for treatment selection (efficacy, safety profile, quality of life, patients preference, physician's preference, comorbidities, other)
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Further Overall Survival parameters
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Best observed tumor response
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Time to progression
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Overall response rate
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Duration of response
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Progression-free-survival
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Disease control rate
Effectiveness of treatment with encorafenib and cetuximab | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Duration of disease control
Patient reported outcomes during treatment with encorafenib plus cetuximab - evaluated with EORTC QLQ C-30 | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  EORTC QLQ C-30 questionnaires (European Organisation for Research and Treatment of Cancer Quality of Life C-30 questionnaires) to assess quality of life of cancer patients; comprises 30 items, 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms. Only in case of prospective inclusion.
Patient's treatment satisfaction - overall | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  4-point scale: very satisfied, satisfied, dissatisfied, very dissatisfied
Physician's treatment satisfaction - differentiated by efficiency, safety and overall | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  4-point scale: very satisfied, satisfied, dissatisfied, very dissatisfied
Safety and tolerability of treatment with encorafenib and cetuximab - Adverse events and adverse reactions including time to onset and time to resolution | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  Number of patients with Adverse Events and maximum grade per patient, Adverse Drug Reactions, Adverse Drug Reactions grade 3/4, Serious Adverse Events, Serious Adverse Drug Reactions
Treatment duration | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  From date to first treatment until date of last treatment (single compounds and whole treatment)
Treatment dose intensity | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  From date to first treatment until date of last treatment (single compounds and whole treatment)
Number of treatment interruptions | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  From date to first treatment until date of last treatment (single compounds and whole treatment)
Duration of treatment interruptions | Through encorafenib plus cetuximab treatment completion, an average of 9 months
  From date to first treatment until date of last treatment (single compounds and whole treatment)

CONTACTS AND LOCATIONS:
Locations (67):
- Austria (4):
  - Clinic, Braunau am Inn, Upper Austria
  - Clinic, Linz, Upper Austria
  - Clinic, Feldkirch, Voralberg
  - Clinic, Vienna
- Germany (63):
  - Practice, Offenburg, Baden-Wurttemberg
  - Medical Care Centre, Ulm, Baden-Wurttemberg
  - Clinic, Ulm, Baden-Wurttemberg
  - Practice, Augsburg, Bavaria
  - Practice, Donauwörth, Bavaria
  - Clinic, Erlangen, Bavaria
  - Practice, München, Bavaria
  - Practice, Würzburg, Bavaria
  - Medical Car Centre, Aschaffenburg, Bayer
  - Medical Care Centre, Potsdam, Brandenburg
  - Practice, Celle, Lower Saxony
  - Medical Care Centre, Goslar, Lower Saxony
  - Practice, Göttingen, Lower Saxony
  - Medical Practice, Hanover, Lower Saxony
  - Practice, Hanover, Lower Saxony
  - Practice, Leer, Lower Saxony
  - Clinic, Weißenfels, Lower Saxony
  - Medical Practice, Wilhelmshaven, Lower Saxony
  - Practice, Rostock, Mecklenburg-Vorpommern
  - Clinic, Rostock, Melcklenburg-Vorpommern
  - Clinic, Aachen, North Rhine-Westphalia
  - Clinic, Bochum, North Rhine-Westphalia
  - Practice, Bonn, North Rhine-Westphalia
  - Clinic, Bonn, North Rhine-Westphalia
  - Practice, Bottrop, North Rhine-Westphalia
  - Clinic, Essen, North Rhine-Westphalia
  - Practice, Moers, North Rhine-Westphalia
  - Medical Care Centre, Mönchengladbach, North Rhine-Westphalia
  - Medical Care Centre, Mülheim, North Rhine-Westphalia
  - Medical Care Centre, Neuss, North Rhine-Westphalia
  - Clinic, Paderborn, North Rhine-Westphalia
  - Medical Care Centre, Porta Westfalica, North Rhine-Westphalia
  - Practice, Stolberg, North Rhine-Westphalia
  - Practice, Troisdorf, North Rhine-Westphalia
  - Clinic, Wuppertal, North Rhine-Westphalia
  - Practice, Bad Kreuznach, Rhineland-Palatinate
  - Practice, Kaiserslautern, Rhineland-Palatinate
  - Practice, Worms, Rhineland-Palatinate
  - Clinic, Saarbrücken, Saarland
  - Practice, Dresden, Saxony
  - Prctice, Naunhof, Saxony
  - Clinic, Torgau, Saxony
  - Practice, Halle, Saxony-Anhalt
  - Clinic, Köthen, Saxony-Anhalt
  - Practice, Köthen, Saxony-Anhalt
  - Clinic, Flensburg, Schleswig-Holstein
  - Clinic, Eisenach, Thuringia
  - Hospital, Aschaffenburg
  - Medical Care Centre, Berlin
  - Practice, Berlin
  - Clinic, Berlin
  - Private Practice, Berlin
  - Private Practice, Dresden
  - Hospital, Esslingen am Neckar
  - Practice, Hamburg
  - Private Practice, Heidelberg
  - Private Practice, Leer
  - Private Practice, Lübeck
  - Private Practice, Naunhof
  - Private Practice, Offenburg
  - Private Practice, Oldenburg in Holstein
  - Private Practice, Schorndorf
  - Private Practice, Würzburg

IPD SHARING:
Plan to Share IPD: No